CLINICAL TRIAL: NCT01515995
Title: Nebulized Magnesium Sulfate Versus Normal Saline as a Vehicle for Albuterol in Children With Moderate to Severe Asthma Exacerbation: a Randomized Controlled Trial
Brief Title: Nebulized Magnesium Sulfate in Children With Moderate to Severe Asthma Exacerbation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ( STU 072011-043)
Record Dates: First submitted 2012-01-11; First posted 2012-01-24 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Magnesium sulfate; Childhood asthma; Emergency department
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulfate group (Experimental): 15 mg albuterol in 22 ml of magnesium sulfate solution (880 mg) via nebulizer over one hour
  Interventions: Drug: Nebulized magnesium sulfate
- Normal Saline group (Active Comparator): 15 mg albuterol in 22 ml of normal saline solution via nebulizer over one hour
  Interventions: Drug: Nebulized magnesium sulfate

INTERVENTIONS:
Drug: Nebulized magnesium sulfate — 15 mg albuterol in 22 ml of magnesium sulfate solution (880 mg) via nebulizer over one hour
  Versus
  15 mg albuterol in 22 ml of normal saline via nebulizer over one hour
  Other Names: Inhaled magnesium sulfate

SUMMARY:
The purpose of this study is to evaluate the effectiveness of nebulized magnesium sulfate as a vehicle for albuterol in children with moderate to severe asthma exacerbation.

DETAILED DESCRIPTION:
Patients presenting to the Emergency Department for acute asthma exacerbation will receive standard care of up to three doses of albuterol and ipratropium bromide plus oral steroid medication. Those seven years of age and older who require further treatment will be screened for eligibility. Eligibility screening will comprise measurement of forced expiratory volume in one second (FEV1) with a bedside spirometer by a respiratory therapist. Children under the age of seven are generally unable to complete spirometry maneuvers and will thus be excluded. The Pediatric Asthma Severity Score (PASS) will also be noted by a respiratory therapist. Patients able to complete spirometry testing and with an FEV1 less than 70% of predicted (the definition of moderate asthma exacerbation) will be enrolled. Enrolled patients will be randomized to receive either Children's Medical Center standard care of 15 mg albuterol diluted in 22 ml of normal saline or the study intervention of 15 mg of albuterol diluted in 22 ml of magnesium sulfate solution. This solution will be prepared at the time of use by a pharmacist in the Emergency Department and will consist of 22 ml of a commercially available 40 mg/ml magnesium sulfate solution (880 mg). The nebulizer treatment will be given over approximately one hour via a large volume nebulizer at 25 ml/hr. Physicians, nurses, and respiratory therapists will be blinded to the diluent used. Vital signs will be noted at baseline. Heart rate, heart rhythm, respiratory rate, and pulse oximetry will be monitored continuously while blood pressure will be measured at baseline and every 15 minutes during study medication administration. The study physician, treating physician, and/or bedside nurse will monitor these values for any clinically significant changes. At the end of the 15 mg albuterol treatment FEV1 and PASS will again be noted. Any further treatments needed, as determined by the treating physician, will be given following Children's Medical Center standard of care. At the discretion of the treating physician intravenous magnesium sulfate may be used post study intervention. The dose used for study participants will be the Children's Medical Center standard dose of 75 mg/kg (max 3 g) minus 880 mg to avoid the risk of magnesium sulfate overdose. Further treatments and patient disposition will be observed by study personnel and noted. Bounce-back rates will be collected by review of enrolled patients' medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ seven years
* Previous diagnosis of asthma or previous episode of wheezing treated with beta-agonist medication
* Able to complete bedside spirometry
* FEV1 < 70% predicted

Exclusion Criteria:

* Known allergy to magnesium sulfate
* Known contra-indication to albuterol
* Respiratory distress occurring as a result of bedside spirometry
* History of neuromuscular disease, cardiac disease, renal disease, or underlying chronic lung disease
* Pregnancy
* Use of oral steroid medication within 72 hours of presentation
* Radiographic evidence of pneumonia at presentation
* Intubation during the current encounter prior to study enrollment
* Administration of intravenous magnesium sulfate prior to study enrollment
* Prior participation in this study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Badawy, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnesium Sulfate Group: 15 mg albuterol in 22 ml of magnesium sulfate solution (880 mg) via nebulizer over one hour
  Nebulized magnesium sulfate: 15 mg albuterol in 22 ml of magnesium sulfate solution (880 mg) via nebulizer over one hour
  Versus
  15 mg albuterol in 22 ml of normal saline via nebulizer over one hour
- Normal Saline Group: 15 mg albuterol in 22 ml of normal saline solution via nebulizer over one hour
  Nebulized magnesium sulfate: 15 mg albuterol in 22 ml of magnesium sulfate solution (880 mg) via nebulizer over one hour
  Versus
  15 mg albuterol in 22 ml of normal saline via nebulizer over one hour
Period: Overall Study
Arm/Group | Magnesium Sulfate Group | Normal Saline Group
Started | 25 | 25
Completed | 22 | 21
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate Group | Normal Saline Group | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 21 | 43
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.8 [7 to 17] | 10.8 [8 to 17] | 10.8 [7 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in One Second (FEV1) %
Description: Change in forced expiratory volume in one second (FEV1) as measured by bedside spirometry before and after study intervention.
Time Frame: Baseline and one hour after treatment
Measure: Mean (95% Confidence Interval); unit: Percentage of FEV1
Arm/Group | Magnesium Sulfate Group | Normal Saline Group
Number analyzed (Participants) | 22 | 21
Percentage of FEV1 | 3.6 [0.9 to 6.3] | 5 [1.7 to 8.4]

ADVERSE EVENTS:
Arm/Group | Magnesium Sulfate Group | Normal Saline Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magnesium Sulfate Group (N=25) | Normal Saline Group (N=25)
Burning sensation in the nose (Respiratory, thoracic and mediastinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes